CLINICAL TRIAL: NCT02628951
Title: Phase II Ramucirumab/Paclitaxel as Second-line Treatment in Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma With Integrative Genomic Analysis
Brief Title: Ramucirumab/Paclitaxel as Second-line Treatment in Metastatic Gastric or Gastroesophageal Junction Adenocarcinoma With Integrative Genomic Analysis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Samsung Medical Center (Other)
Responsible Party: Principal Investigator, Jeeyun Lee, MD,PhD,Division of hematology-oncology,Department of medicine, Samsung Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-11-110
Record Dates: First submitted 2015-12-06; First posted 2015-12-11 (Estimated); Last update posted 2020-11-19 (Actual); Status verified 2020-11

CONDITIONS: Gastric Adenocarcinoma; Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — Ramucirumab; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ramucirumab + Paclitaxel (Experimental): Ramucirumab injection for intravenous (I.V.) use, supplied in single-use 500-mg/50-mL vials containing 10 mg/mL of product in histidine buffer, administered as an I.V. infusion after dilution at 8 mg/kg every 2 weeks in the absence of disease progression, toxicity requiring cessation, or withdrawal for any other reason.
  Paclitaxel will be administered at a dose of 80 mg/m2 on Days 1, 8 and 15 of a 28-day cycle in the absence of disease progression, toxicity requiring cessation, or withdrawal for any other reason.
  Interventions: Drug: Ramucirumab; Drug: Paclitaxel

INTERVENTIONS:
Drug: Ramucirumab — Ramucirumab injection for intravenous (I.V.) use, supplied in single-use 500-mg/50-mL vials containing 10 mg/mL of product in histidine buffer, administered as an I.V. infusion after dilution at 8 mg/kg every 2 weeks in the absence of disease progression, toxicity requiring cessation, or withdrawal for any other reason.
Drug: Paclitaxel — Paclitaxel will be administered at a dose of 80 mg/m2 on Days 1, 8 and 15 of a 28-day cycle in the absence of disease progression, toxicity requiring cessation, or withdrawal for any other reason.

SUMMARY:
Vascular endothelial growth factor is expressed in gastric cancer, and expression has been associated with more aggressive clinical disease. Vascular endothelial growth factor expression has been noted in 51% of gastric cancer specimens in one series (versus no expression in normal epithelium or superficial gastritis). Vascular endothelial growth factor expression in resected gastric cancer is associated with tumor recurrence and shorter survival. Maeda et al. studied 95 gastric cancer patients following resection with curative intent, and noted a significantly shorter survival in 34 patients whose tumor endothelium expressed VEGF (as detected via immunohistochemistry) versus 61 patients without endothelial VEGF expression (p<0.05). Yoshikawa and colleagues observed similar survival differences in resected gastric cancer patients based on levels of circulating (plasma) VEGF at time of resection. Circulating VEGF is significantly higher in gastric cancer patients versus those without neoplasia. Elevated circulating VEGF was also associated with shorter survival in a European cohort undergoing gastric cancer resection; there was no survival beyond 30 months in 24 patients with serum VEGF >533 pg/mL versus a 30-month survival rate >35% for 34 patients with VEGF levels below this threshold (p<0.0001, log-rank test). Recently, Jüttner and colleagues noted reduced survival following R0 resection in gastric cancer patients whose tumors expressed VEGF-C or VEGF-D, with the most robust association between expression and reduced survival for patients whose tumors expressed both VEGF-C and VEGF-D.

Investigational inhibition of VEGF Receptor 2 in gastric cancer xenografts (TMK-1 cell line) is associated with reduced tumor growth. DC101 therapy in this model is associated with significant reductions in tumor vascularity (as measured by CD-31 expression) and increases in endothelial and tumor apoptosis.

The results of the REGARD and RAINBOW studies are consistent with the idea that tumor- related angiogenesis contributes to the pathophysiology of gastric cancer and demonstrate the ability of ramucirumab to represent an improvement in the care of patients with gastric cancer whose disease has progressed after prior chemotherapy.

ELIGIBILITY:
Inclusion Criteria:

1. The patient has histologically or cytologically confirmed gastric carcinoma, including gastric adenocarcinoma or GEJ adenocarcinoma. (Patients with adenocarcinoma of the distal esophagus are eligible if the primary tumor involves the GEJ.)
2. The patient has metastatic disease or locally recurrent, unresectable disease.
3. The patient has measureable or evaluable disease as determined by standard computed tomography (CT) or magnetic resonance imaging (MRI) imaging. Examples of evaluable, nonmeasurable disease include gastric, peritoneal, or mesenteric thickening in areas of known disease, or peritoneal nodules that are too small to be considered measurable by Response Evaluation Criteria in Solid Tumors (RECIST version 1.1) (48).
4. The patient has experienced disease progression during treatment or within 4 months after the last dose of first-line therapy for metastatic disease.

   * Acceptable prior chemotherapy regimens for this protocol are combination chemotherapy regimens that include platinum and/or fluoropyrimidine components (acceptable prior platinum agents are cisplatin, carboplatin, or oxaliplatin; acceptable prior fluoropyrimidine agents are 5-FU, capecitabine, or S-1). Regimens including a third agent, such as an anthracycline or a taxane, are acceptable provided a fluoropyrimidine and/or a platinum were used.
   * Recurrence during or within 6 months of completion of adjuvant chemotherapy (capecitabine, 5-FU, or TS-1) will be considered as first-line chemotherapy.
5. The patient's disease is not amenable to potentially curative resection.
6. The patient is ≥18 years of age.
7. The patient has resolution to Grade ≤1 (or to Grade ≤2 in the case of neuropathy) by the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI- CTCAE), Version 4.03, of all clinically significant toxic effects of prior chemotherapy, surgery, radiotherapy, or hormonal therapy (with the exception of alopecia).
8. The patient has an Eastern Cooperative Oncology Group performance status (ECOG PS) score of 0 or 1.
9. The patient has adequate hepatic function as defined by a total bilirubin ≤1.5 mg/dL (25.65 µmol/L), and aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3.0 times the upper limit of normal (ULN; or 5.0 times the ULN in the setting of liver metastases).
10. The patient does not have:

    * cirrhosis at a level of Child-Pugh B (or worse) or
    * cirrhosis (any degree) and a history of hepatic encephalopathy or clinically meaningful ascites resulting from cirrhosis. Clinically meaningful ascites is defined as ascites from cirrhosis requiring diuretics or paracentesis.
11. The patient has adequate renal function as defined by a serum creatinine ≤1.5 times the ULN, or creatinine clearance (measured via 24-hour urine collection) ≥40 mL/minute (that is, if serum creatinine is >1.5 times the ULN, a 24-hour urine collection to calculate creatinine clearance must be performed).
12. The patient's urinary protein is ≤1+ on dipstick or routine urinalysis (UA; if urine dipstick or routine analysis is ≥2+, a 24-hour urine collection for protein must demonstrate <1000 mg of protein in 24 hours to allow participation in this protocol).
13. The patient has adequate hematologic function, as evidenced by an absolute neutrophil count (ANC) ≥1000/µL, hemoglobin ≥9 g/dL (5.58 mmol/L), and platelets ≥100,000/µL.
14. The patient must have adequate coagulation function as defined by international normalized ratio (INR) ≤1.5 and a partial thromboplastin time (PTT) ≤5 seconds above the ULN (unless receiving anticoagulation therapy). Patients on full-dose anticoagulation must be on a stable dose (minimum duration 14 days) of oral anticoagulant or low molecular weight heparin. If receiving warfarin, the patient must have an INR ≤3.0 and no active bleeding (that is, no bleeding within 14 days prior to first dose of protocol therapy) or pathological condition present that carries a high risk of bleeding (for example, tumor involving major vessels or known varices). Patients on anticoagulation therapy with unresected primary tumors or local tumor recurrence following resection are not eligible.
15. If the patient has received prior anthracycline therapy as part of his or her first-line regimen, the patient is able to engage in ordinary physical activity without significant fatigue or dyspnea (equivalent to New York Heart Association Class I function) (49).
16. Because the teratogenicity of ramucirumab is not known, the patient, if sexually active, must be postmenopausal, surgically sterile, or using effective contraception (hormonal or barrier methods).
17. Female patients of childbearing potential must have a negative serum pregnancy test within 7 days prior to enrollment.
18. The patient is able to provide informed written consent.
19. Feasible biopsy site

Exclusion Criteria:

1. The patient has documented and/or symptomatic brain or leptomeningeal metastases.
2. The patient has experienced any Grade 3 to 4 GI bleeding within 3 months prior to enrollment.
3. The patient has experienced any arterial thromboembolic events, including but not limited to myocardial infarction, transient ischemic attack, cerebrovascular accident, or unstable angina, within 6 months prior to enrollment.
4. The patient has an ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, symptomatic or poorly controlled cardiac arrhythmia, uncontrolled thrombotic or hemorrhagic disorder, or any other serious uncontrolled medical disorders in the opinion of the treating physician.
5. The patient has ongoing or active psychiatric illness or social situation that would limit compliance with treatment.
6. The patient has uncontrolled or poorly controlled hypertension (>160 mmHg systolic or >100 mmHg diastolic for >4 weeks) despite standard medical management.
7. The patient has a serious or nonhealing wound, ulcer, or bone fracture within 28 days prior to enrollment.
8. The patient has received chemotherapy, radiotherapy, immunotherapy, or targeted therapy for gastric cancer within 2 weeks prior to enrollment.
9. The patient has received any investigational therapy within 30 days prior to enrollment.
10. The patient has undergone major surgery within 28 days prior to enrollment, or subcutaneous venous access device placement within 7 days prior to enrollment.
11. The patient has received prior therapy with an agent that directly inhibits VEGF (including bevacizumab), or VEGF Receptor 2 activity, or any antiangiogenic agent.
12. The patient is receiving chronic antiplatelet therapy, including aspirin, nonsteroidal anti- inflammatory drugs (NSAIDs; including ibuprofen, naproxen, and others), dipyridamole or clopidogrel, or similar agents. Once-daily aspirin use (maximum dose 325 mg/day) is permitted.
13. The patient has elective or planned major surgery to be performed during the course of the clinical trial.
14. The patient has a known allergy to any of the treatment components.
15. The patient is pregnant or breastfeeding.
16. The patient is known to be positive for infection with the human immunodeficiency virus (HIV).
17. The patient has known alcohol or drug dependency.
18. The patient has a concurrent active malignancy other than adequately treated nonmelanomatous skin cancer, other noninvasive carcinoma, or in situ neoplasm.
19. The patient has a known hypersensitivity to ramucirumab or any of the excipients.
20. The patient may not have received more than 1 prior therapy in the metastatic setting.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2016-05-26 (Actual); Primary Completion 2019-01-02 (Actual); Study Completion 2019-01-02 (Actual)

PRIMARY OUTCOMES:
objective response rate | every 6weeks
  To evaluate response rate of Ramucirumab in combination with paclitaxel per RECIST 1.1

SECONDARY OUTCOMES:
response rate according to molecular subtypes | through study completion, an average of 1 year
  To analyze the response rate according to molecular subtypes identified through the ACRG effort, with an integrative genomic analysis to identify predictive markers (i.e. angiogenesis signatures) for treatment response

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Kim ST, Sa JK, Oh SY, Kim K, Hong JY, Kang WK, Kim KM, Lee J. Comprehensive molecular characterization of gastric cancer patients from phase II second-line ramucirumab plus paclitaxel therapy trial. Genome Med. 2021 Jan 25;13(1):11. doi: 10.1186/s13073-021-00826-w. PMID 33494793